CLINICAL TRIAL: NCT02959411
Title: Tolvaptan for the Management of Acute Decompensated Heart Failure in Patients With Advanced or Refractory Heart Failure
Brief Title: Tolvaptan for Advanced or Refractory Heart Failure
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low accrual rate
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Jonathan Howlett, Clinical Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB16-0064
Record Dates: First submitted 2016-10-17; First posted 2016-11-09 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Heart Failure; Hyponatremia
MeSH Terms: conditions — Heart Failure; Hyponatremia | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tolvaptan (Experimental): Tolvaptan 15-60 mg, once daily for 4 days or until hospital discharge
  Interventions: Drug: Tolvaptan
- Standard of care diuretic therapy (Active Comparator): Usual standard of care diuretic therapy for patients with acute decompensated heart failure
  Interventions: Drug: Standard of care diuretic therapy

INTERVENTIONS:
Drug: Tolvaptan — Tolvaptan is a selective vasopressin receptor antagonist that inhibits activation of the V2 receptor and synthesis and insertion of the aquaporin2 channel into the apical membrane of the renal collecting duct. Tolvaptan inhibits the reabsorption of free water, inducing free water diuresis and increasing serum sodium levels without adversely influencing electrolyte levels or stimulating the sympathetic nervous system or renin-angiotensin system.
  Other Names: Samsca
  Arms: Tolvaptan
Drug: Standard of care diuretic therapy — Usual standard of care diuretic therapy for patients hospitalized with acute decompensated heart failure
  Arms: Standard of care diuretic therapy

SUMMARY:
This study will clarify the clinical usefulness of Tolvaptan therapy in patients with complicated acute decompensated heart failure and hyponatremia (low blood sodium).

DETAILED DESCRIPTION:
Despite its demonstrated efficacy and tolerability, Tolvaptan remains underutilized for the treatment of acute decompensated heart failure (ADHF) in many centers. Post-hoc analysis suggests that Tolvaptan may provide optimal outcomes in patients with more advanced heart failure (HF) including those with cardiorenal syndrome, marked hyponatremia and severe congestion, or a combination of those conditions. The efficacy of Tolvaptan in HF patients with loop diuretic resistance and in those requiring inotropic support remains uncertain.

The purpose of this study is to examine the benefit of Tolvaptan versus the current standard of care diuretic therapy for patients hospitalized with ADHF and evidence of advanced or complex HF with severe hyponatremia. Patients with advanced or complex disease are defined as those with suboptimal diuretic response over a 48 hour period.

ELIGIBILITY:
Inclusion Criteria:

* Hospital admission for ADHF with volume overload as evidenced by ≥ 2 of the following: Elevated JVP, peripheral edema, ascites, pulmonary rales, congestion on chest X-ray, elevated NT-pro-BNP > 2000 pg/ml
* Inadequate clinical response indicated by body weight loss < 1.0 kg/day over 48 hours despite adequate doses of IV loop diuretic (at least 40 mg furosemide daily) and fluid restriction 2 L/24 hours.
* ≥1 of the following over the preceding 48 hours: Potential need for inotropic support to improve urine output, and/or renal insufficiency (estimated glomerular filtration rate <45 mL/min/1.73 m2)
* Serum sodium ≤134 mmol/L
* ≥18 years-old

Exclusion Criteria:

* Cardiac surgery within 60 days of enrollment
* Planned cardiac mechanical support or transplant; subjects with previously implanted ventricular assist device (VAD) will not be excluded
* Need for intravenous pressor support for symptomatic hypotension
* Biventricular pacemaker placement within the last 60 days
* Hemofiltration or dialysis
* Known cirrhosis
* Supine systolic arterial blood pressure less than 85 mmHg
* Refusal or inability to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-10; Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in body weight | From randomization to 96 hours after randomization

SECONDARY OUTCOMES:
Total 96 hour urine output | From randomization to 96 hours post randomization
  Measured in ml urine
Subjective change in shortness of breath | 48 hours after randomization and 96 hours post randomization
  As assessed by a 5 point Likert scale
Change in renal function | From randomization to 7 days post randomization
  Measured by estimated glomerular filtration rate
Proportion of patients developing worsening renal function (WRF) | From randomization to 7 days post randomization
  Categorical measure- need for renal replacement therapy or ultrafiltration or increase in serum creatinine by > 26 umol/L
Change in serum sodium | From randomization to 7 days post randomization
  Measured in mmol/L
Length of hospitalization | From hospital admission to 30 days post randomization
  Number of days in hospital
Need for intensive care unit admission | From hospital admission to 30 days post randomization
  Categorical measure (yes/no)
Need for positive inotropic agent use | From randomization to 7 days post randomization
  Categorical measure (yes/no)
Composite of Worsening Renal Function or need for inotropic agent | From randomization to 7 days post randomization
  Worsening Renal Function defined as increase from serum creatinine at randomization of more than 30 umol/L at any time from randomization to 7 days. This is a categorical outcome (yes/no)
30 day cardiovascular death and/or hospitalization | From Randomization to 30 days post randomization
  Categorical outcome (yes/no)
Clinical markers of congestion | From randomization to 96 hours after randomization
  Described as total number of the presence of Jugular venous pressure (JVP) level, edema, rales, orthopnea, 3rd heart sound
Change in N-terminal brain natriuretic peptide (NT-pro BNP) | From randomization to 96 hours post randomization compared to baseline
  Measurement calculated in absolute value of NT-pro-BNP

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Howlett, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No